CLINICAL TRIAL: NCT02423746
Title: Assessing and Addressing Behaviors in Children With Hearing Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Matthew Bush, MD, Matthew Bush, MD, Assistant Professor, University of Kentucky, University of Kentucky
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 1012142740-CTSAPilot-Bush
Record Dates: First submitted 2015-03-23; First posted 2015-04-22 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Hearing Loss; Attention Deficit and Disruptive Behavior Disorders; Parenting
MeSH Terms: conditions — Hearing Loss; Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): The control group will include 3 hearing aid (HA) and 3 cochlear implant (CI) caregiver-child dyads.
  Parents in the control group will receive an initial assessment session followed by three behavioral placebo sessions followed by a post-placebo-intervention assessment. All sessions will be delivered in the patients' usual hearing clinics and will last between 60 and 90 minutes. One month post-intervention, participants will complete post-test measures repeating baseline measures, plus acceptability ratings of intervention.
  Interventions: Behavioral: Behavioral Placebo
- Intervention Group (Experimental): The intervention group will include 3 hearing aid (HA) and 3 cochlear implant (CI) caregiver-child dyads.
  Intervention parents receive the initial assessment session followed by the 3-session Family Check Up Behavioral Parenting Training Program (BPT) within one month of baseline assessment followed by a post-intervention assessment. All sessions will be delivered in the patients' usual hearing clinics and will last between 60 and 90 minutes. One month post-intervention, participants will complete post-test measures repeating baseline measures, plus acceptability ratings of intervention.
  Interventions: Behavioral: Family Check Up Behavioral Parenting Training Program (BPT)

INTERVENTIONS:
Behavioral: Family Check Up Behavioral Parenting Training Program (BPT) — The Family Check Up is an evidence-based Behavioral Parenting Training (BPT) program focused on harnessing parents' motivation to change and skills training.
  Intervention parents receive the initial assessment session followed by 3 Family Check-up Sessions within one month of baseline assessment followed by a post-intervention assessment. All sessions will be delivered in the patients' usual hearing clinics and will last between 60 and 90 minutes. One month post-intervention, participants will complete post-test measures repeating baseline measures, plus acceptability ratings of intervention.
  Arms: Intervention Group
Behavioral: Behavioral Placebo — The Behavioral Placebo sessions will consist of presentations of information about healthy lifestyles.
  Parents in the control group will receive an initial assessment session followed by three behavioral placebo sessions followed by a post-placebo-intervention assessment. All sessions will be delivered in the patients' usual hearing clinics and will last between 60 and 90 minutes. One month post-intervention, participants will complete post-test measures repeating baseline measures, plus acceptability ratings of intervention.
  Arms: Control Group

SUMMARY:
Purpose:

This study is a feasibility trial of an existing evidence-based behavioral parent training program with parents of preschool-aged children who were born deaf or hard of hearing (DHH).

The hypotheses of this study are (a) that a randomized control trial of the Family Check Up with this population will be feasible, (b) parents will rate the intervention as acceptable, and (c) a signal of effect will be observable among intervention group parents compared to controls for the following outcome variables: child behaviors, parenting behaviors, and parenting sense of competence.

DETAILED DESCRIPTION:
24 participants, comprising 6 parents and their preschool-aged child with a cochlear implant (CI; n=12) and 6 parents and their preschool-aged child with a hearing aid (HA; n=12) will be identified and recruited at routine clinic visits through university-affiliated hearing clinics. A dyad will consist of the child and his or her primary caregiver. Eligible participants will include children with clinically elevated behavior problems, as determined by having scored between the 70th and 90th percentiles on the Child Behavioral Checklist/1.5-5 (CBCL/1.5-5).

3 HA and 3 CI dyads will be randomized to the intervention group, and 3 HA and 3 CI dyads will be randomized to the control group. The intervention will consist of 3 Family Check-Up sessions within one month of baseline assessment. The control condition will consist of 3 behavioral placebo session within the same time frame, in which general information about healthy lifestyles will be presented. All intervention and control sessions will be delivered in the patients' usual hearing clinics. Each session will last between 60 and 90 minutes. One month post-intervention, all parent participants will complete post-test measures repeating baseline measures, plus acceptability ratings of the intervention.

Feasibility data will be collected via process measures of recruitment, retention, and session attendance. Acceptability will be measured with a parent-completed satisfaction survey. Measures of parenting behaviors, parent self-efficacy, parent-satisfaction, parent competence, child disruptive behaviors, parenting stress, and parental depression will also be piloted in preparation for a future study.

ELIGIBILITY:
Inclusion Criteria:

* Parent is age 18 years or older and the custodial guardian
* The child is aged 3-5 years and lives full-time in the caregiver's home
* The child has had a hearing aid or cochlear implant for at least 6 months and is currently being treated for hearing loss
* The child scores above the 70th but below the 90th percentile on the externalizing subscale of the CBCL/1.5-575 (i.e., elevated level of disruptive behavior problems without clear need for specialized behavioral services)
* Parent can speak, understand, and read English

Exclusion Criteria:

* The child has been diagnosed with a severe developmental condition (e.g., extreme developmental delay, severe autism, or debilitating neurological conditions, for which this intervention may not be adequate or appropriate)
* The parent already has accessed behavioral health services for the child

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of sessions attended by each enrolled parent | 3 months

SECONDARY OUTCOMES:
Ability to recruit 12 parent-child dyas in the allotted time frame | 10 months
COACH fidelity rating form | 10 months months
  Measuring interventionist adherence and competence
Time required per participant to complete all instruments | Up to 3 hours
Proportion of missing data across all instruments and within each instrument | 4 months
Proportions of each full instrument and interview that are successfully completed | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Bush, MD, Principal Investigator — University of Kentucky; Christina R Studts, PhD, Principal Investigator — University of Kentucky
Locations (3):
- United States (3):
  - Lexington Hearing and Speech Academy, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Heuser Hearing Institute, Louisville, Kentucky